CLINICAL TRIAL: NCT01435226
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of GS-5885, GS-9451, Tegobuvir and Ribavirin (RBV) Compared With GS-5885, GS-9451 With Tegobuvir or RBV in Treatment-Experienced Subjects With Chronic Genotype 1a or 1b Hepatitis C Virus (HCV) Infection
Brief Title: GS-5885, GS-9451, Tegobuvir and Ribovirin in Treatment-Experienced Subjects With Chronic Genotype 1a Or 1b Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-248-0131
Record Dates: First submitted 2011-09-13; First posted 2011-09-16 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; Rapid Virologic Response; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; Tegobuvir; Treatment Experienced; HCV RNA; Polymerase inhibitor; Protease inhibitor; Interferon intolerant; Interferon ineligible; GS-9190; GS-9451; GS-5885; Chronic Genotype 1a or 1b
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — ledipasvir; GS-9451; tegobuvir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): GS-5885 90 mg QD + GS-9451 200 mg QD + tegobuvir 30 mg BID + RBV BID
  Interventions: Drug: GS-5885; Drug: GS-9451; Drug: tegobuvir; Drug: Ribavirin
- Arm 2 (Active Comparator): GS-5885 90 mg QD + GS-9451 200 mg QD + tegobuvir 30 mg BID + RBV placebo BID
  Interventions: Drug: GS-5885; Drug: GS-9451; Drug: tegobuvir; Drug: placebo to match RBV
- Arm 3 (Active Comparator): GS-5885 90 mg QD + GS-9451 200 mg QD + tegobuvir placebo BID + RBV BID
  Interventions: Drug: GS-5885; Drug: GS-9451; Drug: placebo to match tegobuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: GS-5885 — Drug: GS-5885 tablet
  GS-5885 tablet, 90 mg, QD
Drug: GS-9451 — Drug: GS-9451 tablet
  GS-9451 tablet, 200 mg QD
Drug: tegobuvir — tegobuvir 30 mg BID
  Arms: Arm 1; Arm 2
Drug: placebo to match tegobuvir — tegobuvir placebo BID
  Arms: Arm 3
Drug: placebo to match RBV — Ribovirin placebo BID
  Arms: Arm 2
Drug: Ribavirin — Ribavirin (Copegus®) BID (1000 mg for subjects weighing < 75 kg and 1200 mg for subjects weighing ≥ 75 kg) divided BID
  Arms: Arm 1; Arm 3

SUMMARY:
This is a Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of GS-5885, GS-9451, Tegobuvir and Ribavirin (RBV) Compared with GS-5885, GS-9451 with Tegobuvir or RBV in Treatment-Experienced Subjects with Chronic Genotype 1a or 1b Hepatitis C Virus (HCV) Infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with chronic HCV infection
* Liver biopsy results ≤ 3 years prior to screening indicating the absence of cirrhosis. Alternatively, a non-invasive procedure conducted within 6 months of screening is permitted in countries where allowed
* Monoinfection with HCV genotype (GT) 1a or 1b
* HCV RNA ≥ 104 IU/mL at screening
* Prior treatment and adherence with one course of pegylated interferon alfa and RBV
* The subject's medical records must include sufficient detail of prior treatment with pegylated interferon alfa and RBV (start/stop dates and viral response) to allow for categorization of prior response as either null, partial, breakthrough or relapse.
* Body mass index (BMI) 18-40 kg/m2 inclusive
* Screening ECG without clinically significant abnormalities and with QTcF interval (QT corrected using Fridericia's formula)

  ≤ 450 msec for males and ≤ 470 msec for females.
* Agree to use two forms of highly effective contraception for the duration of the study and for 7 months after the last dose of study medication. Females of childbearing potential must have a negative pregnancy test at screening and baseline.

Exclusion Criteria:

* Discontinuation of prior treatment with pegylated interferon alfa and RBV due to an adverse event, toxicity reasons or were lost to follow-up
* History of significant cardiac disease
* Exceed criteria delineated in Section 4.2 for laboratory measure thresholds related to leukopenia, neutropenia, anemia, thrombocytopenia, and thyroid stimulating hormone (TSH).
* Diagnosis of autoimmune disease, decompensated liver disease, poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease (COPD), HIV, hepatitis B virus (HBV), hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers), hemoglobinopathy, retinal disease, or are immunosuppressed.
* Current abuse of amphetamines, cocaine, opiates, or alcohol. Methadone use is not allowed, however stable buprenorphine maintenance treatment for ≥ 6 months is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 24 weeks
  To evaluate safety and tolerability of combination therapy with GS-5885, GS-9451, tegobuvir and ribavirin or GS-5885, GS-9451 and tegobuvir or GS-5885, GS-9451 and ribavirin.
  Safety will be assessed during the study through the reporting of adverse events, clinical laboratory tests, physical examinations, vital signs and 12-lead ECGs at various time points during the study.
Antiviral Activity | 24 weeks
  To evaluate the antiviral efficacy as measured by sustained virologic response (SVR, defined as HCV RNA < lower limit of quantitation [LLoQ] 24 weeks post-treatment) of combination therapy with GS-5885, GS-9451, tegobuvir and RBV compared with GS-5885, GS-9451 and tegobuvir or GS-5885, GS-9451 and RBV in treatment-experienced subjects with chronic genotype 1a or 1b HCV infection

SECONDARY OUTCOMES:
Viral Dynamics | 10 days
  To characterize the viral dynamics of GS-5885, GS-9451 and tegobuvir. The median change from baseline in HCV RNA and time-weighted average change from baseline through Day 10 will be assessed based on plasma HCV RNA sampling times to characterize the viral dynamics of GS-5885, GS-9451 and tegobuvir.
Composite (or Profile) of Pharmacokinetics Composite (or Profile) of Pharmacokinetics | predose, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose
  To characterize the steady state pharmacokinetics of GS-5885, GS-9451, tegobuvir and ribavirin (if appropriate). Cmax, Tmax, Clast, Tlast, Ctau, λz, AUCtau and T ½
Antiviral Efficacy | 24-48 weeks
  To evaluate the antiviral efficacy (as defined by SVR) of adding pegylated interferon alfa-2a (PEG) and RBV (Arm 2 only) for 24-48 weeks to the original treatment regimen in subjects who experience viral breakthrough or relapse and enter the Rescue Therapy Substudy

CONTACTS AND LOCATIONS:
Overall Officials: John McNally, PhD, Study Director — Gilead Sciences
Locations (51):
- United States (37):
  - University of Arizona, Tucson, Arizona
  - Advanced Clinical Research Institute, LLC, Anaheim, California
  - California Liver Institute, Beverly Hills, California
  - SCTI Research Foundation Liver Center, Coronado, California
  - University of California, San Diego, La Jolla, California
  - Lightsource Medical, Los Angeles, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Kaiser Permanente, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - San Jose Gastroenterology, San Jose, California
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Avail Clinical Research, LLC, DeLand, Florida
  - University of Miami, Center for Liver Diseases, Miami, Florida
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Weill Medical College of Cornell Univeristy, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Southwest Infectious Disease Clinical Research, Inc, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - The University of Texas Health Sciences Center at Houston, Houston, Texas
  - Alamo Medical Research, Ltd., San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Bon Secours St. Mary's Hospital of Richmond, Inc., Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Germany (14):
  - Leber- and Studienzentrum am Checkpoint, Berlin
  - Charite - Universitatsmedizin Berlin Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt
  - Medizinische Universitatsklinik, Freiburg im Breisgau
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum der Universität Heidelberg, Heidelberg
  - Gastroenterologisch-Hepatologisches Zentrum Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Johannes Gutenberg University Hospital, Mainz
  - Klinikum Innenstadt der LMU Munchen, München
  - Universitätsklinikum Würzburg - Med Klinik und Poliklinik, Würzburg